CLINICAL TRIAL: NCT05277363
Title: A Natural History Study of Surfeit Locus Protein 1 (SURF1)-Associated Leigh Syndrome
Brief Title: A Study of the Natural Course of SURF1 Deficiency
Status: Withdrawn | Type: Observational
Why Stopped: The study stopped early, before enrolling its first participant
Sponsor: Taysha Gene Therapies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TSHA-104-RG-001
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Leigh Syndrome
Keywords: SURF1-associated Leigh Syndrome; Biomarkers; Epidemiology study; Genotype-phenotype correlation data; Leigh Syndrome; Primary Mitochondrial Disease; SURF1 deficiency; Natural History study; Neurodegenerative disease
MeSH Terms: conditions — Leigh Disease; Neurodegenerative Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum/Plasma/Cerebrospinal fluid (CSF) biobanking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective cohort: Parents/caregivers of participants with SURF1 deficiency will provide information regarding diagnosis, onset of symptoms, and course of the disease and participants will be assessed prospectively over time using standardized qualitative and quantitative tools.
  Interventions: Other: None (Observational study)

INTERVENTIONS:
Other: None (Observational study) — No investigational intervention, marketed product, or placebo will be administered to study participants in this study.
  Other Names: Observational study

SUMMARY:
The purpose of the study is to prospectively and systematically collect standardized clinical information, to describe important features of the disease course of SURF1 deficiency. These include but are not limited to symptomatology, clinical course, and risk factors for severe disease and complications.

DETAILED DESCRIPTION:
Participant eligibility for the study will be determined during a screening period lasting up to 45 days. In-clinic follow visits will occur over several days every 6 months for 2 years from baseline. Thereafter, annual telephone follow-up contact will be conducted for 2 additional years. Thus, the active study duration for each participant will be up to approximately 2 years and the total duration per participant will be approximately 4 years.

The study will be conducted in the United States and select sites outside the United States based on incidence data.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent/assent provided by the participant based on participant's cognitive ability as determined by Principal Investigator (PI), and/or participant's parent(s) or legally authorized representative(s).
* Participant is < 18 years of age at time of initial informed consent.
* Displays one or more clinical features consistent with SURF1 deficiency, including but not limited to, hypotonia, motor delays, motor regression, failure to thrive, language delays, and/or language regression.
* Genetic diagnosis of SURF1 pathogenic or likely pathogenic mutation(s), either compound heterozygous or homozygous mutations. If variants are of uncertain significance (VUS), verify documentation of cytochrome c oxidase (COX) activity deficiency.
* Ability to travel to the study site and adhere to study-related follow-up examinations and/or procedures and provide access to participant's medical records.

Exclusion Criteria:

* Any known genetic abnormality (other than SURF1 deficiency), including but not limited to a chromosomal aberration or molecularly known or clinically suspected progressive neurometabolic disorder or dementia, that confounds the clinical phenotype.
* The presence of significant non-SURF1-related central nervous system (CNS) impairment/behavioral disturbances that would confound the scientific rigor or interpretation of results of the study or a known history of perinatal asphyxia, kernicterus, carbon monoxide or methanol intoxication.
* Current participation in a therapeutic study or participation in a therapeutic study within 30 days prior to enrollment in the present study.
* Prior or current treatment with gene or stem cell therapy.
* Any condition that, in the opinion of the Site Investigator, could put the participant at undue risk and/or would ultimately prevent the completion of study procedures.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants with SURF1 deficiency
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Newcastle Paediatric Mitochondrial Disease Scale (NPMDS) | From baseline until follow-up (up to 24 months/early termination)
  The NPMDS is scored by section (domain), and the final (total) score is the sum of all section scores. Function is rated over preceding 4-week period, according to participant and/or caregiver. NPMDS is subdivided by patient age (0-24 months, 2-11 years, and 12-18 years).

SECONDARY OUTCOMES:
Change from baseline in Head Control Scale | From baseline until follow-up (up to 24 months/early termination)
  Head control will be evaluated using the Head Control Scale (which ranges 0 to 16, with 0 representing no function and 4 representing normal function in each of the 4 domains).
Change from baseline in Gross Motor Function Measure (GMFM) | From baseline until follow-up (up to 24 months/early termination)
  The Gross Motor Function Measure will measure the child's capacity for gross motor function. Scores are based on a 0 to 100% scale with higher percentage indicating better function.
Change from baseline in Vineland Adaptive Behavior Scales Third Edition (Vineland-3) | From baseline until follow-up (up to 24 months/early termination)
  Vineland-3 forms aid in diagnosing and classifying intellectual and developmental disabilities and other disorders. The individual's overall adaptive functioning is described by a total score and three subdomain scores. The scores ranges from 20 to 140, with higher numbers indicating better performance.

CONTACTS AND LOCATIONS:
Locations (1):
- UTSW Medical Center at Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No